CLINICAL TRIAL: NCT04958967
Title: A Phase Ib Open-Label, Randomization Multi-Center Study to Evaluate Efficacy and Safety of FURMONERTINIB MESILATE in PATIENTS with LOCALLY ADVANCED or METASTATIC NON-SMALL CELL LUNG CANCER HARBOURING EGFR EXON 20 INSERTION MUTATION
Brief Title: Phase Ib Study of FURMONERTINIB in Patients with NSCLC Having Exon 20 Insertion Mutation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The protocol need to review
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALSC015AST2818
Record Dates: First submitted 2021-07-05; First posted 2021-07-12 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2021-07

CONDITIONS: NSCLC
MeSH Terms: interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treated subjects will receive Furmonertinib 240mg/day, (Experimental): treated subjects will receive Furmonertinib 240mg/day, QD, PO, under fasted state, until progressive disease, death or intolerability.
  Interventions: Drug: Furmonertinib 240mg
- treated subjects will receive Furmonertinib 160mg/day (Experimental): treated subjects will receive Furmonertinib 160 mg/day, QD, PO, under fasted state, until progressive disease, death or intolerability.
  Interventions: Drug: Furmonertinib 160mg

INTERVENTIONS:
Drug: Furmonertinib 240mg — treated subjects will receive Furmonertinib 240mg/day
  Arms: treated subjects will receive Furmonertinib 240mg/day,
Drug: Furmonertinib 160mg — treated subjects will receive Furmonertinib 160mg/day
  Arms: treated subjects will receive Furmonertinib 160mg/day

SUMMARY:
This is a phase 1 multi-center clinical study. To explore the efficacy and safety of Furmonertinib Mesilate at different doses in locally advanced or metastatic NSCLC patients with EGFR exon 20 insertion mutation.

The study plans to enroll 20subjects, including 20 treated patients aThe subjects will receive Furmonertinib Mesilate 240 mg/day or 160mg/day until disease progression, death or intolerability.

The primary endpoint is Overall Response Rate (ORR) as Assessed by the Independent Review Committee (IRC); the secondary study endpoints include ORR（ Assessed by the Investigator），DCR，DOR，DpR，PFS，OS，CNS ORR（ Assessed by the Independent Review Committee） In addition, the peripheral blood ctDNA will be collected and analyzed in this study

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged ≥18 years;
* Histologically or cytopathologically confirmed primary non-small cell lung cancer (NSCLC) with predominant non-squamous cell histology;
* Treated patients: progress or intolerance after receiving at least one and no more than three lines of systemic treatment (including at least one chemotherapy or immunotherapy) for locally advanced or metastatic NSCLC disease; If the completion time of adjuvant or neoadjuvant treatment is less than or equal to 6 months from the time of the first disease progression, it is evaluated in accordance with the criteria for treated patients Treatment-naïve patients t without any systemic anti-tumor therapy for locally advanced or metastatic NSCLC; If the completion time of adjuvant or neoadjuvant treatment is more than 6 months from the time of first disease progression, the patients be eligible for enrollment to the study;
* The Participants should provide enough ctDNA in peripheral blood during the screening period, and at the same time, they should provide enough advanced tumor tissue sections as far as possible for central laboratory testing to confirm the mutation type of EGFR 20 exon (please refer to the manual of central laboratory for details);
* Participants meeting either of the following conditions (in accordance with the AJCC 8th edition TNM stage classification for lung cancer):
* Having at least one measurable lesion (in accordance with RECIST1.1). Note: measurable lesion can neither be subject to local therapy as radiotherapy nor used for biopsy in screening period; if there is only one measurable lesion, this lesion will be permitted to be biopsied. However, the baseline radiological examination can be performed for this lesion at least 14 days after biopsy.
* Adequate organ function as shown in the laboratory test, including: 1)Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; platelet count (PLT) ≥ 100 × 109/L; hemoglobin (HGB) ≥ 90 g/L; 2)Serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), AST and ALT ≤ 2.5 × ULN (total bilirubin ≤ 3 × ULN, AST and ALT ≤ 5 × ULN in patients with hepatic metastasis); 3)Creatinine clearance (CrCL) ≥ 50 ml/min (using Cockcroft- Gault formula); Prothrombin time (PT) ≤ 1.5 × ULN;
* ECOG PS score 0-1 at screening, no obvious exacerbation of disease within 2 weeks prior to screening;
* Life expectancy >12 weeks after the first dose of investigational product;
* Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of investigational product; female subjects of non-childbearing potential may not undergo pregnancy test or contraception. Non-childbearing potential is defined as: 50 years and above, no use of hormone therapy and amenorrhea for at least 12 months; or having received sterilization operation. Female subjects at childbearing age and male subjects agree to take effective contraceptive measures during the study and within 6 months after drug discontinuation;
* Being able to understand and voluntarily participate in the study, and sign the informed consent form.

Exclusion Criteria：

Any potential participant who meets any of the following criteria will be excluded fromparticipating in the study:

* NSCLC with predominant squamous cell histology, small cell lung cancer or neuroendocrine carcinoma indicated by Histology or cytology test;
* Expected to receive other anti-tumor therapy other than the investigational product during the study;
* Treated patients: having previously received systematic anti-tumor therapy with 3rd-generation EGFR TKI (marketed drugs or drugs under development) ;

  1）Therapeutic drugs (such as dzd9008, tak788, jnj-372, bocitinib, etc.) for EGFR 20 exon insertion mutation; 2)The third generation of EGFR TKI (marketed or in research drug); 3） The first and second generation EGFR TKI (marketed drugs or drugs in Research) targeting the insertion mutation of EGFR 20 exon had objective remission;
* Having received the following therapies:

  1. Having been irradiated for >30% bone marrow or a large area within 4 weeks prior to the first dose of investigational product;
  2. Having received major surgery within 4 weeks prior to the first dose of investigational product or plan to receive major surgery during the study with exception of the surgical procedures to establish vascular access, biopsy through mediastinoscopy or thoracoscopy;
  3. Use of a potent CYP3A4 inhibitor within 7 days prior to the first dose of investigational product or a potent CYP3A4 inducer within 21 days prior to the first dose of investigational product;
  4. use of the traditional Chinese medicine or traditional Chinese medicine preparation with tumor indication, or traditional Chinese medicine or traditional Chinese medicine preparation with adjuvant anti-tumor effect within two weeks prior to the first dose of investigational product or expected to be required during the study;
* Having participated in the clinical trial and received the investigational product or device within 4 weeks or at least 5 half-lives prior to the first dose of investigational product;
* Having received other anti-tumor drugs within 14 days prior to the first dose of investigational product;
* Concurrent spinal cord compression or symptomatic brain metastasis. Subjects with stable brain metastasis will be eligible. Stable brain metastasis is defined as the patients who have completed regular treatment for brain metastasis, are clinically stable or asymptomatic for at least two weeks and do not need steroid therapy. If the investigator considers there is no indication of immediate radical treatment, patients with asymptomatic brain metastasis will be eligible.
* The toxicity caused by previous anti-tumor therapy has not recovered to ≤CTCAE grade 1 (CTCAE 5.0) ( except alopecia, sequelae of previous platinum-related neurotoxicity) or the level specified in the inclusion/exclusion criteria;
* Unstable pleural effusion or peritoneal effusion with obvious symptoms; those with stable clinical symptoms for at least 14 days after drainage of pleural effusion or ascites will be eligible;
* Having a history of other malignant tumor, or other concurrent malignant tumors (except those that have undergone radical operation and have no recurrence within 5 years post operation, e.g., cervical carcinoma in situ, basal cell carcinoma of skin and papillary thyroid carcinoma);
* Previous interstitial lung disease (ILD), drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy; or having the clinical manifestations of suspected interstitial lung disease;
* Having severe or uncontrolled systemic disease requiring treatment that is considered by investigators as ineligible for the study, including hypertension, diabetes, chronic heart failure (NYHA Functional Classification III-IV), unstable angina pectoris, myocardial infarction within one year, active hemorrhagic disease, etc.;
* Left ventricular ejection fraction (LVEF) <50% on echocardiography;
* Clinically significant prolonged QT interval or other arrhythmia or clinical status considered by investigators that may increase the risk of prolonged QT interval; for example, QTc>470 ms on ECG at resting state, complete left bundle branch block, degree III atrioventricular block, congenital long QT syndrome, serious hypokalemia, or current use of drugs that may lead to prolonged QT interval;
* Serious gastrointestinal dysfunction, or disease that may affect the intake, transportation or absorption of investigational product;
* Known hepatitis B virus (positive HBsAg), hepatitis C virus (positive HCV Ab) or human immunodeficiency virus (positive HIV antibody) infection;
* Infectious disease requiring intravenous medication;
* Known history of mental disease or drug abuse, and currently having an attack or still taking drugs;
* Known or suspected allergy to Furmonertinib or other components of its preparation;
* Female subjects or female partners of male subjects who are pregnant or lactating, or plan to be pregnant during the study;
* Poor compliance, inability to comply with the study procedures, restriction or requirements;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
ORR, objective response rate | up to 12 months
  IRC assessed objective response rate (ORR) using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 in participants with epidermal growth factor receptor EGFRmutations. These outcome is based on the visual assessment of tumor size in morphological images provided by computed tomography (CT) or magnetic resonance imaging.ORR is defined as the percentage of participants achieving complete response (CR) and partial response (PR) per RECIST version 1.1. CR: Disappearance of all extranodal target lesions; PR: At least a 30% decrease in Sum of the Longest Diameters (SLD) of target lesions, taking as a reference the baseline SLD.

SECONDARY OUTCOMES:
Duration of Response (DOR) | up to 2 years
  Duration of response is defined as the time interval from the time that the measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that PD is objectively documented.
Disease Control Rate (DCR) | up to 2 years
  DCR is defined as the percentage of participants who have achieved CR, PR, or stable disease (SD) (in the case of SD, measurements must have met the SD criteria at least once after study entry at a minimum interval of 42 days) after the initiation of study drug.
Progression Free Survival (PFS) | up to 2 years
  PFS is defined as the time interval from the date of randomization until the first date at which the criteria for progressive disease (PD) according to RECIST version 1.1 are met or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No